CLINICAL TRIAL: NCT06110650
Title: A Single-arm, Single-center, Exploratory Phase II Study of Surufatinib in Patients With Soft Tissue Sarcoma Who Have Failed Anthracycline-containing Chemotherapy and Who Have Been Successfully Targeted With Antivascular Agents
Brief Title: A Study of Surufatinib in the Treatment of Advanced Soft Tissue Sarcoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Deputy chief of medical oncology, chief physician，Fudan University Shanghai Cancer Center, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2306276-6
Record Dates: First submitted 2023-10-17; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Soft Tissue Sarcoma Adult
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surufatinib (Experimental): surufatinib 300mg orally, once a day, every 21 days for one cycle, treatment until disease progression or intolerance
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Surufatinib 300mg orally, once a day, every 21 days for one cycle, treatment until disease progression or intolerance

SUMMARY:
This is a single-center, open, single-arm, phase II clinical study to investigate the efficacy and safety of patients with soft tissue sarcoma who have failed anthracycline-containing chemotherapy and whose antivascular agents have been effective and failed.

Progression-free survival (PFS) was used as the primary outcome measure to preliminatively estimate the efficacy and safety of 29 patients with soft tissue sarcoma who had failed chemotherapy with anthracyclines and who had received effective and failed antivascular agents. Sofantinib 300mg orally, once a day, with continuous administration every 21 days, until the disease progresses or becomes intolerable; Imaging methods were used every 6 weeks (±7 days) after enrollment according to RECIST1.1 standard to evaluate the efficacy of tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood the study and voluntarily signed the informed consent;
2. Age ≥18 years old;
3. Histologically or cytologically confirmed patients with unresectable or metastatic soft tissue sarcoma;
4. The patient must have at least one measurable lesion (RECIST1.1);
5. Previous failure of anthracycline-containing chemotherapy was defined as disease progression during treatment or within 3 months after the last treatment, or disease progression during adjuvant treatment with anthracycline-containing chemotherapy or within 6 months after adjuvant treatment, and toxic side effects of anthracycline-containing chemotherapy were not tolerated. (Neoadjuvant or adjuvant chemotherapy is allowed in the early stage. If disease progression/recurrence occurs during neoadjuvant/adjuvant therapy or within 6 months after the end of treatment, neoadjuvant/adjuvant therapy is considered a failure of first-line systemic chemotherapy for progressive disease);
6. Patients with previous anti-angiogenic efficacy and failure were defined as: tumor progression occurred in SD or above patients after withdrawal of SD (CR/PR) during the course of anti-angiogenic therapy (including anti-angiogenic small molecule inhibitors or monoclonal antibodies), or tumor progression occurred in SD patients over 12 weeks; Or the toxic side effects of treatment are intolerable.
7. ECOG physical status 0 or 1 points (PS0-2 points for amputees);
8. Expected survival ≥12 weeks;
9. Blood test (without blood transfusion within 14 days)

1) Neutrophil absolute value ≥1.5×10^9/L, platelets ≥100×10^9/L, hemoglobin concentration ≥9g/dL);

2) Liver function test (aspartate aminotransferase and glutamic aminotransferase ≤2.5×ULN, total bilirubin ≤1.5×ULN; In case of liver metastasis, AST and ALT≤5×ULN);

3) Renal function (serum creatinine ≤1.5×ULN, creatinine clearance (CCr)≥60ml/min)

10. Fertile male or female patients voluntarily used effective contraceptive methods, such as double barrier methods, condoms, oral or injectable contraceptives, intrauterine devices, etc., during the study period and within 6 months of the last study dose. All female patients will be considered fertile unless they have undergone natural menopause, artificial menopause, or sterilization (such as hysterectomy, bilateral adnexectomy, or irradiation of radioactive ovaries).

Exclusion Criteria:

1. Patients who have received previous treatment with Surufatinib;
2. Consider toxic reactions associated with anti-vascular targeting drugs if they have previously been intolerable
3. Participated in other domestic unapproved or unmarketed drug clinical trials and accepted the corresponding experimental drug treatment within 4 weeks before enrollment;
4. Received any surgery or invasive treatment or operation (except intravenous catheterization, puncture drainage, etc.) within 4 weeks before enrollment;
5. International Standardized Ratio (INR)>1.5 or partially activated prohemase time (APTT)>1.5×ULN;
6. The investigator identified clinically significant electrolyte abnormalities;
7. The patient currently has high blood pressure that cannot be controlled by drugs, which is defined as: systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg;
8. Unsatisfactory blood glucose control (FBG > 10mmol/L);
9. The patient has any current disease or condition that affects the absorption of the drug, or the patient cannot take sofantinib orally;
10. The patient currently has gastrointestinal diseases such as active gastric and duodenal ulcers, ulcerative colitis, or active bleeding from unresectosed tumors, or other conditions determined by researchers that may cause gastrointestinal bleeding or perforation;
11. Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding within 3 months >30mL, hematemesis, stool, stool blood), hemoptysis (within 4 weeks >5mL of fresh blood) or had a thromboembolic event (including stroke events and/or transient ischemic attacks) within 12 months;
12. Clinically significant cardiovascular disease, including but not limited to the following: acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment; Congestive Heart Failure New York Heart Association (NYHA) Grades > Lv.2; Ventricular arrhythmias requiring medical treatment; LVEF(Left ventricular Ejection Fraction)<50%;
13. Have had other malignancies within the past 5 years, except basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;
14. Active or uncontrolled severe infection;

1) Known human immunodeficiency virus (HIV) infection;

2) A known history of clinically significant liver disease, including viral hepatitis A known hepatitis B virus (HBV) carrier must rule out active HBV infection, i.e., positive HBVDNA (>1×10^4 copies /mL or >2000IU/ml);

3) Known hepatitis C virus infection (HCV) and HCVRNA positive (>1×10^3 copies /mL), or other hepatitis, cirrhosis;

15. The patient has current central nervous system (CNS) metastases or previous brain metastases;

16. Patients with persistent toxicity due to any previous antitumor therapy that has not returned to ≤ grade 2, but with alopecia or lymphocytopenia of any grade are admitted to this study;

17. Women who are pregnant (positive pregnancy test before medication) or breastfeeding;

18. Any other medical condition, a clinically significant metabolic abnormality, abnormal physical examination, or abnormal laboratory examination, which, in the investigator's judgment, reasonably suspects the patient to have a medical condition or condition that is not suitable for the use of the investigational drug (such as the presence of epileptic seizures requiring treatment), or which would affect the interpretation of the study results, or place the patient at a high risk;

19. Urine routine indicated urinary protein ≥2+, and 24-hour urinary protein quantification > 1.0g.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-11-28 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
PFS | PFS is defined as approximately 12 months from the date of enrollment until the date of first recorded progress or the date of death from any cause, whichever comes first
  progression-free survival

SECONDARY OUTCOMES:
ORR | From date of enrollment until the end of treatment or the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Objective Response Rate
OS | OS From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Overall Survival
DCR | From date of enrollment until the end of treatment or the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Disease Control Rate

IPD SHARING:
Plan to Share IPD: No